CLINICAL TRIAL: NCT00422617
Title: Evaluate the Efficacy and Safety of One Course of Amevive in Taiwan Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uni-Pharma (Industry)
Collaborators: Biogen (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: ASIA-7002
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Last update posted 2007-01-17 (Estimated); Status verified 2004-09

CONDITIONS: Chronic Plaque Psoriasis
Keywords: psoriasis; alefacept
MeSH Terms: conditions — Psoriasis | interventions — Alefacept

INTERVENTIONS:
Drug: Alefacept (Amevive)

SUMMARY:
An open-label, multicentre study to evaluate the efficacy and safety of one course of weekly intramuscular administration of Amevive in Taiwan patients with chronic plaque psoriasis

DETAILED DESCRIPTION:
The purpose of the present study is to establish the efficacy and safety of one course of once weekly 15 mg intramuscular (IM) administration of AMEVIVE in an alternate study population and to address the issue of peak time to response by measuring the proportion of patients achieving a ≥ 75% reduction in PASI at any time after completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent
* Must be >= 16 years of age
* Must have been diagnosed with chronic plaque psoriasis at least one year and require systemic or phototherapy
* Must have CD4+ lymphocyte count at or above the lower limit of normal
* Must have a BSA >= 10%

Exclusion Criteria:

* Current erythrodermic, generalized pustular, or guttate psoriasis
* Serious local infection or systemic infection within 3 months prior to the first dose of alefacept
* History of any clinical significant disease that would be contraindicated for this study as determined by the investigator
* Prior history of systemic malignancy, untreated localised skin canceer or a >10 squamous cell carcinoma
* Current enrollment in any other investigational drug study within 30 days prior to study drug administration
* Treatment with systemic immunosuppressant agents within the 4 weeks prior to study drug administration.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2005-01; Study Completion 2005-11

PRIMARY OUTCOMES:
To determine TRR75 of one course of once weekly 15 mg intramuscular (IM) administration of AMEVIVE

SECONDARY OUTCOMES:
To determine TRR50, Quality of Life (QOL), the safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Po-Han Huang, Principal Investigator — CGMH